CLINICAL TRIAL: NCT03992456
Title: PULSE: A Randomized, Phase II Open Label Study of PanitUmumab RechaLlenge Versus Standard Therapy After Progression on Anti-EGFR Therapy in Patients With Metastatic and/or Unresectable RAS Wild-Type Colorectal Cancer
Brief Title: Panitumumab, Regorafenib, or TAS-102, in Treating Patients With Metastatic and/or Unresectable RAS Wild-Type Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-GI-1623; NCI-2019-03306 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-GI-1623 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Colon Adenocarcinoma; Metastatic Colorectal Carcinoma; Metastatic Rectal Adenocarcinoma; Stage III Colon Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Colon Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Colon Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Colon Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8; Stage IV Colon Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8; Stage IVA Colon Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Rectal Cancer AJCC v8; Stage IVB Colon Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Rectal Cancer AJCC v8; Stage IVC Colon Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8; Stage IVC Rectal Cancer AJCC v8; Unresectable Colon Adenocarcinoma; Unresectable Colorectal Carcinoma; Unresectable Rectal Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms | interventions — Panitumumab; regorafenib; Trifluridine; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A (panitumumab) (Experimental): Patients receive panitumumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Panitumumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (regorafenib, trifluridine and tipiracil hydrochloride) (Active Comparator): Patients receive trifluridine and tipiracil hydrochloride PO BID on days 1-5 and 8-12, or regorafenib PO QD on days 1-21, at the discretion of the treating physician. Treatment repeats every 28 days for a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Regorafenib; Drug: Trifluridine and Tipiracil Hydrochloride

INTERVENTIONS:
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; E7.6.3; Human IgG2K Monoclonal Antibody; MoAb ABX-EGF; MoAb E7.6.3; Monoclonal Antibody ABX-EGF; Monoclonal Antibody E7.6.3; Vectibix
  Arms: Arm A (panitumumab)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506; Regorafenib Anhydrous
  Arms: Arm B (regorafenib, trifluridine and tipiracil hydrochloride)
Drug: Trifluridine and Tipiracil Hydrochloride — Given PO
  Other Names: Lonsurf; TAS 102; TAS-102; Tipiracil Hydrochloride Mixture with Trifluridine; Trifluridine/Tipiracil; Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102
  Arms: Arm B (regorafenib, trifluridine and tipiracil hydrochloride)

SUMMARY:
This phase II trial studies how well retreatment with panitumumab works compared to standard of care regorafenib or trifluridine and tipiracil hydrochloride (TAS-102) in treating patients with colorectal cancer that is negative for RAS wild-type colorectal cancer has spread to other places in the body (metastatic), and/or cannot be removed by surgery (unresectable), and is negative for resistance mutations in blood. Treatment with panitumumab may interfere with the ability of tumor cells to grow and spread. Some tumors need growth factors to keep growing. Growth factor antagonists, such as regorafenib, may interfere with the growth factor and stop the tumor from growing. Drugs used in chemotherapy, such as TAS-102, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving panitumumab may work better in treating patients with colorectal cancer than with the usual treatment of regorafenib or TAS-102.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the overall survival (OS) in molecularly selected patients with metastatic colorectal cancer (CRC) receiving panitumumab rechallenge versus standard therapy (TAS-102 or regorafenib).

SECONDARY OBJECTIVES:

I. To compare the progression free survival (PFS) in molecularly selected patients with metastatic CRC receiving panitumumab rechallenge versus standard therapy (TAS-102 or regorafenib).

II. To define the objective response rate (ORR) in patients receiving panitumumab rechallenge versus standard therapy (TAS-102 or regorafenib).

III. To define the clinical benefit rate (CBR = complete response + partial response + stable disease >= 4 months) in patients receiving panitumumab rechallenge versus standard therapy (TAS-102 or regorafenib).

IV. To compare the safety and tolerability of panitumumab rechallenge versus standard therapy (TAS-102 or regorafenib).

V. To compare quality of life (QOL) between panitumumab rechallenge versus standard therapy (TAS-102 or regorafenib) as measured by the linear analogue self-assessment (LASA) questionnaires.

CORRELATIVE RESEARCH OBJECTIVES:

I. To assess plasma pharmacodynamics biomarkers of response and resistance to therapy.

II. To explore any correlation between tissue and blood based biomarkers and clinical outcomes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive panitumumab intravenously (IV) over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive trifluridine and tipiracil hydrochloride orally (PO) twice daily (BID) on days 1-5 and 8-12, or regorafenib PO once daily (QD) on days 1-21, at the discretion of the treating physician. Treatment repeats every 28 days for a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 3 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Most recent Guardant360 blood collection date =< 90 days prior to randomization.

  * NOTE: If a patient does not have Guardant360 test results available, enrollment in ACCRU_GI-1611 (COLOMATE) is strongly encouraged.
* Greater than 90 days has elapsed between the most recent treatment with an anti-epidermal growth factor receptor gene (EGFR) therapy (cetuximab or panitumumab) and blood collection for Guardant360 assay.
* Age >= 18 years.
* Histologically and/or cytologically confirmed adenocarcinoma of the colon or rectum that is metastatic and/ or unresectable.
* Documented wild-type in KRAS and NRAS (codons 12, 13, 59, 61, 117, and 146) and in BRAF codon 600, based on tumor tissue taken from primary or metastatic site prior to receipt of anti EGFR therapy.
* Progression, intolerance, or contraindication to:

  * A fluoropyrimidine (e.g., 5-fluorouracil or capecitabine)
  * Oxaliplatin
  * Irinotecan
  * An anti-vascular endothelial growth factor (VEGF) monoclonal antibody (including but not limited to bevacizumab, ramucirumab, or aflibercept).
  * If the tumor has deficient mismatch repair proteins (dMMR) or is microsatellite instability (MSI)-high based on tumor tissue testing, an anti-programmed death (PD)-1 monoclonal antibody (including but not limited to nivolumab or pembrolizumab).
* Clinical or radiographic progression after treatment with an anti-EGFR monoclonal antibody (cetuximab and/or panitumumab) for at least 3 months (minimum of 6 biweekly treatments or 12 weekly treatments at full or partial dose).

  * NOTE: Treatments do not need to be administered consecutively.
  * NOTE: Dose reductions or delays are permitted.
* At least one site of disease that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) criteria that has not been previously irradiated; if the patient has had previous radiation to the target lesion(s), there must be evidence of progression since the radiation.
* Life expectancy >= 3 months per estimation of investigator.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1, or 2.
* Absolute neutrophil count (ANC) >= 1500/mm^3 without colony stimulating factor support (obtained =< 7 days prior to randomization).
* Platelet count >= 75,000 /mm^3 (obtained =< 7 days prior to randomization).
* Hemoglobin > 8.0 g/dL (obtained =< 7 days prior to randomization).
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 7 days prior to randomization).
* Aspartate transaminase (AST) =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer) (obtained =< 7 days prior to randomization).
* Alanine aminotransferase (ALT) =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer) (obtained =< 7 days prior to randomization).
* Calculated creatinine clearance must be > 30 ml/min using the Cockcroft-Gault formula or serum creatinine < 1.5 x ULN (obtained =< 7 days prior to randomization).
* Women of child bearing potential and male partners of women of child bearing potential must agree to use two medically accepted methods of contraception, one of them being a barrier method during the study and for 2 months after the last dose of study drug(s).
* Negative serum pregnancy test done =< 7 days prior to randomization, for women of childbearing potential only.

  * NOTE: Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Postmenopause is defined as amenorrhea >= 12 consecutive months.
  * NOTE: Women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, ovarian suppression or any other reversible treatment.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Capable of understanding and complying with the protocol requirements and has signed the informed consent document.
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study).
* Willing to provide tissue and blood samples for correlative research purposes.
* Willing to allow transfer of tissue and blood samples, clinical information, and outcome data collected from this trial for future research.

Exclusion Criteria:

* Radiation therapy, hormonal therapy, biologic therapy, experimental therapy, or chemotherapy for cancer < 21 days prior to randomization.
* Therapeutic anticoagulation with Vitamin-K antagonists (e.g., warfarin).
* Maximum mutant allele frequency (highest allele frequency reported for any gene mutation) (MAF) less than 0.5% by Guardant360 assay.
* Detection of at least one of the following gene mutation(s) or amplification(s) by Guardant360 assay.

  * BRAFV600E mutation (mutant allele frequency (MAF) >= 0.5% or amplification.
  * EGFR mutation (MAF >= 0.5%). Note: EGFR S492R, K467, and R451C mutations are not an exclusion.
  * ERBB2 (HER2) amplification.
  * KRAS mutation (MAF >= 0.5%) or amplification.
  * MET amplification.
  * NRAS mutation (MAF >= 0.5%) or amplification.
* Prior treatment with both TAS-102 and regorafenib (prior treatment with either TAS-102 or regorafenib is permitted).
* Unable to swallow oral tablets (crushing of study treatment tablets is not allowed).
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens. Note: This includes impaired heart function or clinically significant heart disease.
* Not recovered to baseline or Common Terminology for Adverse Events (CTCAE) version (v)5.0 =< grade 1 from toxicity due to all prior therapies except alopecia, oxaliplatin-related neuropathy, asymptomatic electrolyte abnormalities, and other non-clinically significant adverse events.
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women.
  * Nursing women.
  * Men or women of childbearing potential who are unwilling to employ adequate contraception.
* Patients with known central nervous system (CNS) metastases. Note: Patients with radiated or resected lesions are permitted, provided the lesions are fully treated and inactive (based on repeat imaging >= 30 days after completion of definitive treatment), patients are asymptomatic, and no steroids to control symptoms related to CNS metastases have been administered for at least 30 days.
* Major surgical procedure, open biopsy, or significant traumatic injury =< 28 days prior to randomization (=< 56 days for hepatectomy, open thoracotomy, major neurosurgery) or anticipation of need for major surgical procedure during the course of the study.
* Serious, non-healing wound, ulcer, or bone fracture.
* History of stroke (cerebrovascular accident), transient ischemic attack (TIA), myocardial infarction (MI), unstable angina, cardiac or other vascular stenting, angioplasty, or cardiac surgery =< 6 months prior to randomization.
* History of cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers, calcium channel blockers, or digoxin =< 6 months prior to randomization.
* Known history of congestive heart failure - New York Heart Association (NYHA) >= class II.
* Known history of human immunodeficiency virus (HIV) seropositivity, acute or chronic active hepatitis B or C infection, or other serious chronic infection requiring ongoing treatment.
* History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest computed tomography (CT) scan.
* Subjects with any previously untreated or concurrent cancer that is distinct in primary site or histology from colorectal cancer except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor. Note: Subjects surviving a cancer that was curatively treated and without evidence of disease or biochemical relapse (undetectable PSA for prostate cancer) for 3 or more years before randomization are allowed. All cancer treatments must be completed at least 3 years prior to randomization.
* Uncontrolled hypertension (systolic pressure > 150 mm HG or diastolic pressure > 90 mm Hg [National Cancer Institute (NCI)-CTCAE v5.0]) on repeated measurement despite optimal medical management.
* Evidence or history of bleeding diathesis or coagulopathy.
* Any hemorrhage or bleeding event >= NCI CTCAE v5.0 grade 3, =< 4 weeks prior to randomization.
* Ongoing active infection > grade 2 NCI-CTCAE v5.0.
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulation given during the course of this trial.

  * EXCEPTION: Cetuximab
* Any known history of malabsorption condition.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
* Use of any herbal remedy (e.g. St. John's wort) =< 7 days prior to randomization.
* Use of strong CYP3A4 inducers or inhibitors =< 7 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-10-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John H Strickler, Principal Investigator — Academic and Community Cancer Research United
Locations (18):
- United States (18):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Panitumumab): Patients receive panitumumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity.>
  > Panitumumab: Given IV>
  > Quality-of-Life Assessment: Ancillary studies>
  > Questionnaire Administration: Ancillary studies
- Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride): Patients receive trifluridine and tipiracil hydrochloride PO BID on days 1-5 and 8-12, or regorafenib PO QD on days 1-21, at the discretion of the treating physician. Treatment repeats every 28 days for a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity.> > Quality-of-Life Assessment: Ancillary studies>
  > Questionnaire Administration: Ancillary studies>
  > Regorafenib: Given PO>
  > Trifluridine and Tipiracil Hydrochloride: Given PO
Period: Overall Study
Arm/Group | Arm A (Panitumumab) | Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride)
Started | 5 | 6
Completed | 0 | 0
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disease progression | 4 | 5
Not completed — Emergency surgery unrelated to treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Panitumumab) | Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride) | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (11.17) | 64.0 (6.75) | 62.8 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (8.82) | 24.1 (4.57) | 25.8 (6.72)
Primary Tumor Site [Count of Participants; unit: Participants]
  Left | 5 | 5 | 10
  Right | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the Time from randomization to death from any cause. The distribution of overall survival will be estimated using the method of Kaplan-Meier. Overall survival will be compared between the 2 treatment arms using the un-stratified log-rank test will be used.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A (Panitumumab): Patients receive panitumumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity.
  >
  > Panitumumab: Given IV
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
- Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride): Patients receive trifluridine and tipiracil hydrochloride PO BID on days 1-5 and 8-12, or regorafenib PO QD on days 1-21, at the discretion of the treating physician. Treatment repeats every 28 days for a maximum of 24 cycles in the absence of disease progression or unacceptable toxicity.
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
  >
  > Regorafenib: Given PO
  >
  > Trifluridine and Tipiracil Hydrochloride: Given PO
Arm/Group | Arm A (Panitumumab) | Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride)
Number analyzed (Participants) | 5 | 6
months | 7.5 [7.2 to NA] — Due to an insufficient number of participants with events, the upper confidence interval was not able to be estimated | 8.3 [4.9 to NA] — Due to an insufficient number of participants with events, the upper confidence interval was not able to be estimated
Statistical Analysis 1: Comparison: Arm A (Panitumumab) vs Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride); Test type: Superiority; p = 0.5126, Un-Stratified Log-rank

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to documentation of disease progression or death due to any cause, whichever is first. If the patient did not have any disease evaluation post randomization, PFS will be censored at one day after randomization. The distribution of progression free survival will be estimated using the method of Kaplan-Meier. Progression free survival will be compared between the 2 treatment arms using the log-rank test which is used for the primary endpoint analysis.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Panitumumab) | Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride)
Number analyzed (Participants) | 5 | 6
months | 5.1 [2.0 to NA] — Due to an insufficient number of participants with events, the upper confidence interval was not able to be estimated | 3.7 [2.0 to NA] — Due to an insufficient number of participants with events, the upper confidence interval was not able to be estimated
Statistical Analysis 1: Comparison: Arm A (Panitumumab) vs Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride); Test type: Superiority; p = 0.1512, Un-Stratified Log-rank

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Defined as the number of patients with a complete response (CR) or partial response (PR) (as defined by the Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) divided by the number of evaluable patients in each arm. ORR will be compared between the 2 treatment arms. Confidence intervals for the true success proportion will be calculated according to the approach of Clopper and Pearson.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Arm A (Panitumumab) | Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride)
Number analyzed (Participants) | 5 | 6
percent | 20.0 [0.51 to 71.6] | 0.0 [0.0 to 45.93]
Statistical Analysis 1: Comparison: Arm A (Panitumumab) vs Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride); Test type: Superiority; p = 0.2506, Chi-squared

4. Secondary Outcome: Clinical Benefit Rate
Description: Defined as the number of patients with a complete response (CR), partial response (PR), or stable disease for >= 4 months (as defined by the RECIST 1.1) divided by the number of evaluable patients in each arm. Confidence intervals for the true success proportion will be calculated according to the approach of Clopper and Pearson.
Time Frame: 4 months
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Arm A (Panitumumab) | Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride)
Number analyzed (Participants) | 5 | 6
percent | 20.0 [0.51 to 71.6] | 16.67 [0.42 to 64.12]
Statistical Analysis 1: Comparison: Arm A (Panitumumab) vs Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride); Test type: Superiority; p = 0.8865, Chi-squared

5. Secondary Outcome: Incidence of Adverse Events
Description: The maximum grade for each type of adverse event will be recorded for each patient in each cycle. The number of patients experiencing grade 3 or higher adverse events will be compared using Chi-Square or Fisher's Exact tests.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Panitumumab) | Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride)
Number analyzed (Participants) | 5 | 6
Participants | 1 | 3
Statistical Analysis 1: Comparison: Arm A (Panitumumab) vs Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride); Test type: Superiority; p = 0.5455, Fisher Exact

6. Secondary Outcome: Patient-reported Quality of Life
Description: Patients reported quality of life (QOL) outcomes will be collected using the Linear Analog Self-Assessment (LASA) Questionnaire. Data will be collected each cycle. Mean values of the first question (regarding overall QOL) at each cycle will be plotted, and stratified by arm. Additional analyses using data collected from the LASA questionnaire may be performed. Score from 0-10, 0 is worse and 10 is better.
Time Frame: 2 years
Population: This analysis was not conducted due to no patient response rates.
Arm/Group | Arm A (Panitumumab) | Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride)
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Cell Free Tumor Deoxyribonucleic Acid (cfDNA)
Description: A report will be generated for each clinical specimen, which may include (but not limited to) the presence or absence of relevant gene mutations or amplifications, along with the allele frequency. Mutations of interest include KRAS and NRAS exons 2, 3, and 4, BRAF, PIK3CA, EGFR, AKT, PTEN, MAP2K1, and MET. Amplifications of interest include MET, EGFR, KRAS, and ERBB2. Genes and alterations analyzed will be based on best available science at the time of analysis.
Time Frame: Baseline, at restaging, and at disease progression
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Circulating Protein Studies
Description: Plasma samples will be analyzed for multiple soluble protein analytes, which may include (but not limited to) HGF, c-MET, EGF, HBEGF, TGF-alpha, EGFR, HER2, and CD73.
Time Frame: Up to 3 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Tumor Tissue Studies
Description: Comprehensive mutational analysis will be performed on archived formalin fixed paraffin embedded (FFPE) tumor samples. This analysis may include, but is not limited to Next Generation Sequencing (NGS) and IHC where appropriate.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Arm A (Panitumumab) | Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 5/5 | 5/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 2/6
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Panitumumab) (N=5) | Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride) (N=6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Panitumumab) (N=5) | Arm B (Regorafenib, Trifluridine and Tipiracil Hydrochloride) (N=6)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (12) | 4 (12)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 3 (3)
Weight loss (Investigations) | 0 (0) | 2 (3)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (17) | 1 (2)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT03992456/Prot_SAP_000.pdf